CLINICAL TRIAL: NCT06118411
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy, Safety, and Tolerability of Upadacitinib in Adult and Adolescent Subjects With Non-Segmental Vitiligo Who Are Eligible for Systemic Therapy
Brief Title: A Study To Assess Adverse Events and Effectiveness of Upadacitinib Oral Tablets in Adult and Adolescent Participants With Vitiligo
Acronym: Viti-Up
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-044; 2023-506195-27-00 (Other: EU CT)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo
Keywords: Vitiligo; Non-Segmented Vitiligo; Viti-Up; Upadacitinib
MeSH Terms: conditions — Vitiligo | interventions — upadacitinib; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Study 1, Period A: Group 1 (Experimental): Participants will receive upadacitinib 15 mg once daily for 48 weeks.
  Interventions: Drug: Upadacitinib
- Study 1, Period A: Group 2 (Placebo Comparator): Participants will receive placebo once daily for 48 weeks.
  Interventions: Drug: Placebo
- Study 2, Period A: Group 1 (Experimental): Participants will receive upadacitinib 15 mg once daily for 48 weeks.
  Interventions: Drug: Upadacitinib
- Study 2, Period A: Group 2 (Placebo Comparator): Participants will receive placebo once daily for 48 weeks.
  Interventions: Drug: Placebo
- Study 1, Period B: Group 1 Open-Label Extension Period (Experimental): Participants that were randomized to receive upadacitinib in Period A Group 1, will continue to receive upadacitinib 15 mg once daily for 112 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Study 1, Period B: Group 2 Open-Label Extension Period (Experimental): Participants that were randomized to receive placebo in Period A Group 2, will receive upadacitinib 15 mg once daily for 112 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Study 2, Period B: Group 1 Open-Label Extension Period (Experimental): Participants that were randomized to receive upadacitinib in Period A Group 1, will continue to receive upadacitinib 15 mg once daily for 112 weeks in Period B.
  Interventions: Drug: Upadacitinib
- Study 2, Period B: Group 2 Open-Label Extension Period (Experimental): Participants that were randomized to receive placebo in Period A Group 2, will receive upadacitinib 15 mg once daily for 112 weeks in Period B.
  Interventions: Drug: Upadacitinib
- (Optional) Study 3, Period B: Open Label Upadacitinib (Experimental): Open Label Upadacitinib Participants will receive upadacitinib 15 mg once daily for 112 weeks
  Interventions: Drug: Upadacitinib; Other: NB-UVB (narrow-band ultraviolet B) Phototherapy
- (Optional) Study 3: (Experimental): Participants will receive 15 mg upadacitinib once daily for 112 weeks and NB-UVB for up to 28 weeks
  Interventions: Drug: Upadacitinib; Other: NB-UVB (narrow-band ultraviolet B) Phototherapy

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Other Names: ABT-494; Rinvoq
  Arms: (Optional) Study 3, Period B: Open Label Upadacitinib; (Optional) Study 3:; Study 1, Period A: Group 1; Study 1, Period B: Group 1 Open-Label Extension Period; Study 1, Period B: Group 2 Open-Label Extension Period; Study 2, Period A: Group 1; Study 2, Period B: Group 1 Open-Label Extension Period; Study 2, Period B: Group 2 Open-Label Extension Period
Drug: Placebo — Oral Tablets
  Arms: Study 1, Period A: Group 2; Study 2, Period A: Group 2
Other: NB-UVB (narrow-band ultraviolet B) Phototherapy — NB-UVB phototherapy is a commonly used treatment modality in participants with vitiligo and can be administered in an office setting or at home 2 times per week
  Arms: (Optional) Study 3, Period B: Open Label Upadacitinib; (Optional) Study 3:

SUMMARY:
Vitiligo is a common chronic autoimmune disease that causes the body's immune system to attack its own pigment producing skin cells. This study is to evaluate how safe and effective upadacitinib is in participants with non-segmental vitiligo (NSV). Adverse effects and change in disease activity will be assessed.

Upadacitinib is an approved drug for various immune-mediated inflammatory diseases and is currently being investigated for the treatment of NSV. There will be 2 replicate studies running at the same time (Study 1 and Study 2 with periods A and B) and an optional exploratory Narrow-Band Ultraviolet B (NB-UVB) phototherapy study (Study 3). In Period A, participants are placed in 1 of 2 groups called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will receive placebo and 2 in 3 chance participants will receive upadacitinib. In Period B, all participants will receive upadacitinib. Approximately 270 adult and adolescent participants with NSV will be enrolled in each main study ((Study 1 and Study 2, 540 subjects total) at approximately 90 sites worldwide with an option for adult participants who completed Period A of either study and did not achieve T-VASI 90 at week 48 while on study drug, to enter Study 3.

In Studies 1 and 2: Period A, participants will receive oral tablets of upadacitinib or placebo once a day for 48 weeks. In Period B, participants will receive oral tablets of upadacitinib 15 mg once a day for 112 weeks. Participants will be followed up for 30 days. Study 3 participants will receive upadacitinib monotherapy or upadacitinib with NB-UBV phototherapy for at least 24 weeks followed by upadacitinib alone.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of non-segmented vitiligo (NSV).
* At Screening and Baseline Visits, participants must satisfy at least 1 of the following criteria:

  * >= 0.5 F-VASI and 5 <= T-VASI < 50 AND have failed at least 1 topical corticosteroid and/or at least 1 topical calcineurin inhibitor for vitiligo; or
  * >= 0.5 F-VASI and 5 <= T-VASI < 50 AND have a sign of actively progressing vitiligo; or
  * >= 0.5 F-VASI and 10 <= T-VASI < 50.

Exclusion Criteria:

* Segmental or localized vitiligo.
* History of active skin disease other than vitiligo that could interfere with the assessment of vitiligo.
* >33% leukotrichia in areas of vitiligo on the face or > 33% leukotrichia in areas of vitiligo on the body (including the face).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Total Vitiligo Area Scoring Index (T-VASI) 50 (≥ 50% Improvement in T-VASI From Baseline) | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100.
Percentage of Participants Achieving Facial-Vitiligo Area Scoring Index (F-VASI) 75 (≥ 75% Improvement in F-VASI From Baseline) | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.

SECONDARY OUTCOMES:
Percentage of Participants Achieving F-VASI 50 (≥ 50% Improvement in F-VASI From Baseline) | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.
Percentage of Participants Achieving F-VASI 75 (≥ 75% Improvement in F-VASI From Baseline) | Week 24
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.
Percent Change from Baseline in F-VASI | Week 24
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.
Percent Change From Baseline in T-VASI | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100.
Percentage of Participants Achieving F-VASI 90 (≥ 90% Improvement in F-VASI From Baseline) | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.
Percentage of Participants Achieving T-VASI 75 (≥ 75% Improvement in T-VASI From Baseline) | Week 48
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100.
Percentage of Participants Achieving 3D Imaging Facial Vitiligo 40 (≥ 40% Reduction in Facial Vitiligo Area Measured by 3D Digital Imaging from Baseline) (Study 1 Only) | Week 48
  3D imaging will be used to objectively quantify the facial vitiligo area.
EU/EMA Only: Percentage of Participants Achieving a Physician's Global Impression of Change - Vitiligo (PhGIC-V) of "Much better (1)" | At Week 48
  The physician rates the overall change in the patients vitiligo by comparing the severity of vitiligo right now with the severity of vitiligo since the subject started the study treatment. Responses range from 1 = "Much better" to 5 = "Much worse."
EU/EMA Only: Percentage of Participants Achieving a Vitiligo Noticeability Scale (VNS) score of "A lot less noticeable (4)" or "No longer noticeable (5)" | At Week 48
  The VNS is a single-item, validated questionnaire used in clinical trials to assess the noticeability of vitiligo lesions following therapy. The item is scored on a 5-point scale: 1 = more noticeable; 2 = as noticeable; 3 = slightly less noticeable; 4 = a lot less noticeable; and 5 = no longer noticeable. A score of 4 or 5 represents treatment success
EU/EMA Only: Percentage of Participants Achieving a Patient's Global Impression of Change-Vitiligo (PaGIC-V) of "Much better (1)" | At Week 48
  The PaGIC-V asks participants to rate the overall change in their vitiligo by comparing the severity of their vitiligo right now with the severity of their vitiligo since they started the study treatment. Responses range from 1 = "Much better" to 5 = "Much worse."

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (148):
- United States (46):
  - Advanced Research Associates - Glendale /ID# 259915, Glendale, Arizona
  - Alliance Dermatology and Mohs Center /ID# 259926, Phoenix, Arizona
  - Private Practice - Dr. Tooraj Raoof /ID# 260055, Encino, California
  - University of California Irvine /ID# 260080, Irvine, California
  - Vitiligo & Pigmentation Institute of Southern California /ID# 259970, Los Angeles, California
  - Dermatology Research Associates /ID# 260056, Los Angeles, California
  - Duplicate_Stanford University /ID# 260081, Redwood City, California
  - Integrative Skin Science and Research /ID# 260060, Sacramento, California
  - University of California Davis Health /ID# 260062, Sacramento, California
  - Clinical Trials Research Institute /ID# 259910, Thousand Oaks, California
  - Skin Care Research Boca Raton /ID# 260094, Boca Raton, Florida
  - Apex Clinical Trials /ID# 260096, Brandon, Florida
  - Florida Academic Dermatology Center /ID# 259919, Coral Gables, Florida
  - Direct Helpers Research Center /ID# 259932, Hialeah, Florida
  - Skin Care Research - Hollywood /ID# 260101, Hollywood, Florida
  - Encore Medical Research /ID# 259963, Hollywood, Florida
  - GSI Clinical Research, LLC /ID# 259918, Margate, Florida
  - Life Clinical Trials /ID# 260097, Margate, Florida
  - Savin Medical Group, LLC /ID# 259968, Miami Lakes, Florida
  - Advanced Clinical Research Institute /ID# 260058, Tampa, Florida
  - Encore Medical Research - Weston /ID# 260542, Weston, Florida
  - Cleaver Medical Group Dermatology /ID# 259925, Dawsonville, Georgia
  - DeNova Research /ID# 260611, Chicago, Illinois
  - Indiana University Health University Hospital /ID# 259974, Indianapolis, Indiana
  - Dawes Fretzin, LLC /ID# 260068, Indianapolis, Indiana
  - Tufts Medical Center /ID# 260088, Boston, Massachusetts
  - UMass Memorial Medical Center /ID# 259921, Worcester, Massachusetts
  - Oakland Hills Dermatology /ID# 260602, Auburn Hills, Michigan
  - Great Lakes Research Group - Bay City /ID# 260600, Bay City, Michigan
  - Hamzavi Dermatology - Canton /ID# 260545, Canton, Michigan
  - Clarkston Dermatology /ID# 260069, Clarkston, Michigan
  - Henry Ford Medical Center - New Center One /ID# 260059, Detroit, Michigan
  - Minnesota Clinical Study Center /ID# 260154, New Brighton, Minnesota
  - Vivida Dermatology- Flamingo /ID# 260609, Las Vegas, Nevada
  - Schweiger Dermatology, P.C. /ID# 260152, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 259909, New York, New York
  - DermResearchCenter of New York, Inc. /ID# 259906, Stony Brook, New York
  - ClinOhio Research Services /ID# 260300, Columbus, Ohio
  - Oregon Medical Research Center /ID# 259911, Portland, Oregon
  - Oregon Dermatology and Research Center /ID# 259917, Portland, Oregon
  - Medical University of South Carolina /ID# 259916, Charleston, South Carolina
  - Bellaire Dermatology Associates /ID# 260044, Bellaire, Texas
  - Dermatology Treatment and Research Center /ID# 260078, Dallas, Texas
  - Innovative Dermatology - Plano /ID# 260628, Plano, Texas
  - Dermatology Clinical Research Center of San Antonio /ID# 260047, San Antonio, Texas
  - Progressive Clinical Research /ID# 260070, San Antonio, Texas
- Argentina (6):
  - Buenos Aires Skin /ID# 259885, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia /ID# 259888, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Psoriahue Med Interdisciplinar /ID# 259890, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto De Investigaciones Clínicas Córdoba /ID# 260371, Córdoba, Córdoba Province
  - Sanatorio 9 de Julio /ID# 260245, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC) /ID# 259889, Buenos Aires
- Belgium (4):
  - Cliniques Universitaires UCL Saint-Luc /ID# 259429, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Les Viviers /ID# 259437, Charleroi, Hainaut
  - UZ Gent /ID# 259430, Ghent, Oost-Vlaanderen
  - CHU de Liege /ID# 259427, Liège
- Bulgaria (4):
  - Ambulatory for Specialized Medical Care-IPSMC-skin and venereal diseases /ID# 259955, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 259956, Sofiya, Sofia
  - Diagnosis - Consult Centre 20 - Sofia /ID# 259953, Sofiya, Sofia
  - Medical Center Cordis /ID# 259954, Pleven
- Canada (8):
  - Dermatology Research Institute - Blackfoot Trail /ID# 261175, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 260239, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 260236, Winnipeg, Manitoba
  - Brunswick Dermatology Center /ID# 260237, Fredericton, New Brunswick
  - LEADER Research /ID# 260407, Hamilton, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 260406, Waterloo, Ontario
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 260241, Québec, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 260238, Saint-Jérôme, Quebec
- China (15):
  - Beijing Tongren Hospital Affiliated To Capital Medical University /ID# 260919, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University /ID# 260136, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University /ID# 259929, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University /ID# 260477, Wuhan, Hubei
  - Second Affiliated Hospital of Xian Jiaotong University /ID# 260011, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University /ID# 260340, Xi'an, Shaanxi
  - Shandong Dermatological Hospital /ID# 260338, Jinan, Shandong
  - Huashan Hospital, Fudan University /ID# 259823, Shanghai, Shanghai Municipality
  - Chengdu Second Municipal People's Hospital /ID# 260423, Chengdu, Sichuan
  - West China Hospital, Sichuan University /ID# 260624, Chengdu, Sichuan
  - Tianjin Medical University General Hospital /ID# 259812, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University /ID# 260017, Kunming, Yunnan
  - Hangzhou Third People'S Hospital /ID# 261005, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 260626, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 259822, Wenzhou, Zhejiang
- France (5):
  - Chu de Nice-Hopital L'Archet Ii /Id# 259442, Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Saint-Andre /ID# 259443, Bordeaux, Gironde
  - CHU Toulouse - Hopital Larrey /ID# 259445, Toulouse, Haute-Garonne
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 259446, Créteil, Paris
  - HCL - Hopital Edouard Herriot /ID# 259444, Lyon, Rhone
- Germany (11):
  - Universitaetsklinikum Erlangen /ID# 260153, Erlangen, Bavaria
  - Klinikum rechts der Isar /ID# 260291, Munich, Bavaria
  - Dermatologie Mahlow /ID# 260148, Blankenfelde-Mahlow, Brandenburg
  - MVZ Dermatologisches Zentrum Bonn GmbH /ID# 260287, Bonn, Hesse
  - Universitaetsklinikum Frankfurt /ID# 260288, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim /ID# 260293, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Muenster /ID# 260147, Münster, North Rhine-Westphalia
  - Universitaetsmedizin Mainz /ID# 260151, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 260289, Dresden, Saxony
  - Private Practice - Dr. Abdou Zarzour /ID# 260290, Halle, Saxony-Anhalt
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 260294, Berlin
- DERMA-B Egeszsegugyi es Szolgaltato - Debrecen - Gyepusor Utca /ID# 260072, Debrecen, Hungary
- Israel (5):
  - Hadassah Medical Center-Hebrew University /ID# 259849, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 259851, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 259850, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 259852, Haifa
  - Rabin Medical Center /ID# 260420, Petah Tikva
- Italy (2):
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Dermatologico San Gallicano /ID# 259771, Rome, Roma
  - ASST degli Spedali Civili di Brescia /ID# 259772, Brescia
- Japan (7):
  - Nagoya City University Hospital /ID# 260551, Nagoya, Aichi-ken
  - Dermatology and Ophthalmology Kume Clinic /ID# 260555, Sakai-shi, Osaka
  - The University of Osaka Hospital /ID# 261285, Suita-shi, Osaka
  - Nippon Medical School Hospital /ID# 260550, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 260552, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 260553, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital /ID# 260554, Kofu, Yamanashi
- Netherlands (3):
  - Bravis Ziekenhuis /ID# 259501, Bergen op Zoom, North Brabant
  - Amphia Ziekenhuis /ID# 259696, Breda, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 259676, Amsterdam, North Holland
- Poland (10):
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski /ID# 259690, Osielsko, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno Badawczy /ID# 260016, Krakow, Lesser Poland Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 259686, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne /ID# 261424, Krakow, Lesser Poland Voivodeship
  - Klinika Osipowicz & Turkowski sp.z.o.o /ID# 259761, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia /ID# 260018, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 259691, Warsaw, Masovian Voivodeship
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik /ID# 259753, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Angelius Provita /ID# 259752, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM /ID# 259757, Szczecin, West Pomeranian Voivodeship
- Portugal (4):
  - Unidade Local de Saude de Coimbra, EPE /ID# 259793, Coimbra
  - Unidade Local de Saude da Regiao de Leiria, EPE /ID# 259789, Leiria
  - Hospital CUF Descobertas /ID# 259788, Lisbon
  - Unidade Local de Saude de Santo Antonio, E.P.E. /ID# 259791, Porto
- Puerto Rico (3):
  - Santa Cruz Behavioral (SCB) Research Center /ID# 260100, Bayamón
  - Dr. Samuel Sanchez PSC /ID# 260090, Caguas
  - Mindful Medical Research /ID# 260092, San Juan
- Slovakia (2):
  - Derma therapy spol /ID# 260838, Bratislava, Bratislava Region
  - Fakultna nemocnica Trnava /ID# 260164, Trnava
- South Korea (5):
  - Chungnam National University Hospital /ID# 260917, Daejeon, Daejeon Gwang Yeogsi
  - Soon Chun Hyang University Hospital Bucheon /ID# 260836, Bucheon-si, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 260880, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 260916, Suwon, Gyeonggido
  - Kyung Hee University Hospital at Gangdong /ID# 260879, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol /ID# 259371, Badalona, Barcelona
  - Hospital Universitario de Getafe /ID# 259376, Getafe, Madrid
  - Hospital Universitario Quironsalud Madrid /ID# 259377, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Clinico San Cecilio /ID# 259374, Granada
  - Grupo Pedro Jaen /ID# 259375, Madrid
  - Consorci Hospital General Universitario de Valencia /ID# 259372, Valencia
  - Hospital Clinico Universitario Lozano Blesa /ID# 259373, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-044